CLINICAL TRIAL: NCT02002195
Title: Modified Folinic Acid-Fluorouracil-Oxaliplatin (FOLFOX) Followed by Capecitabine as First-line Chemotherapy for Elderly or Frail Patients With Metastatic or Recurrent Gastric Cancer
Brief Title: Modified Folinic Acid-Fluorouracil-Oxaliplatin Regimen + Capecitabine for Elderly With Metastatic Gastric Cancer
Acronym: MATURE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Group of Endovascular Oncology (Other)
Responsible Party: Principal Investigator, Vincenzo Catalano, Dr., International Group of Endovascular Oncology
Other Study IDs: MATURE01; MATURE (Other: IGEVO)
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Gastric Cancer
Keywords: metastatic gastric cancer,; elderly,; folinic acid,; fluorouracil,; oxaliplatin,; capecitabine,; overall survival,; progression free survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — Folfox protocol; Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- modified folfox: Oxaliplatin 85 mg/m2 in 2 hours intravenous infusion, + S-leucovorin 200 mg/m2, + 5-FU 2,400 mg/m2 as a 46 hours continuous infusion. The cycles are repeated every 2 weeks for a total of 8 cycle, if tumor response is stable disease, partial or complete response, then maintenance with Capecitabine 1,000 mg twice a day will be administered until disease progression, unacceptable toxicity or treatment refusal by the patient.
  Interventions: Drug: FOLFOX; Drug: Capecitabine

INTERVENTIONS:
Drug: FOLFOX — Oxaliplatin 85 mg/m2 is given as a 2 hours intravenous infusion, concomitant to and S-leucovorin 200 mg/m2, and followed by 5-FU 2,400 mg/m2 as a 46 hours continuous infusion.
  Other Names: oxaliplatin+leucovorin+ 5 Fluorouracil
Drug: Capecitabine — Capecitabine 1,000 mg twice a day will be administered until disease progression, unacceptable toxicity or treatment refusal by the patient.
  Other Names: Xeloda

SUMMARY:
Elderly patients are generally underrepresented in the study populations of combination chemotherapy trials. In gastric cancer patients, oxaliplatin has shown a more favorable toxicity profile than cisplatin. A combination chemotherapy of 5-fluorouracil (5-FU) with oxaliplatin, mainly FOLFOX regimens, has been investigated in numerous phase II studies, using different doses and schedules, and has shown considerable antitumor activity. Insofar as toxicity is concerned, significant toxicities, including myelo-suppression and peripheral neuropathy, are a major issue for elderly patients. A modified FOLFOX regimen by omitting the administration of bolus 5-fluorouracil have shown a good profile of activity and tolerability in the elder population. This study evaluates the efficacy and safety of a modified FOLFOX (m FOLFOX) regimen for up to 8 cycles followed by capecitabine maintenance in elderly patients with metastatic gastric cancer and presenting associated disease(s)

DETAILED DESCRIPTION:
Although the number of deaths from gastric cancer has declined during the past, a large proportion of elderly patients are primarily affected by the disease. The definition of an elderly patient varies according to social and economic situations. However, in most developed and developing countries, 65 or 70 years of age is a commonly used limit because of the decreased role of the subject in the community and society.

Elderly cancer patients often suffer multiple comorbidities, take many medications, and have age-associated physiological problems, such as impaired organ function and functional changes, that make the selection of optimal treatment difficult. This aspect is also hampered by the underrepresentation of older patients in cancer clinical trials. Elderly patients who fulfill the inclusion criteria of clinical trials could experience the same advantages and toxicities from chemotherapy as younger patients. In contrast to physicians' perceptions, older patients do not recognize their age as an important issue for refusing trials [4]. Furthermore, performance status is not helpful to estimate the general condition of elderly patients, and other factors regarding their functional, social, and mental status should be considered [5].

Although the majority of gastric cancer patients are elderly, patients older than 65-70 years have been often excluded from, or underrepresented in, the study populations of combination chemotherapy trials.

There is, moreover, a lack of prospective studies directly comparing the outcomes and the tolerability of chemotherapy in young and elderly patients, although some data are available in gastric cancer from a retrospective analysis . Trumper et al. evaluated retrospectively 1,080 patients who were enrolled into three randomized controlled trias assessing 5-FU-based combination chemotherapy. They found that elderly patients obtained similar benefits from palliative chemotherapy in terms of symptomatic response, tumor regression, and survival, without increased toxicities.

In gastric cancer patients, oxaliplatin has shown a more favorable toxicity profile than cisplatin . A combination chemotherapy of 5-FU with oxaliplatin, mainly FOLFOX regimens, has been investigated in numerous phase II studies, using different doses and schedules, and has shown considerable antitumor activity. Insofar as toxicity is concerned, significant toxicities, including myelo-suppression and peripheral neuropathy, are a major issue for elderly patients. When compared to standard FOLFOX schedules, both weekly and biweekly reduced-dose combinations of oxaliplatin/5- FU without 5-FU bolus showed a more favorable toxicity profile with lower rates of peripheral neuropathy and myelosuppression.

For the palliative treatment of metastatic gastric cancer, a doublet containing oxaliplatin and fluoropyrimidines could be considered as an option. Results from a prospective randomized trial showed the non-inferiority of oxaliplatin, as compared to cisplatin, in the treatment of advanced gastric cancer, while decreasing toxicity. Of interest, a subgroup analysis from a phase III randomized trial reported significantly better results for elderly patients treated with oxaliplatin as compared to cisplatin. In this trial, patients with advanced gastric cancer were randomized to receive a 5-FU-based regimen with cisplatin (FLP regimen) or oxaliplatin (FLO regimen). The primary endpoint of the study, PFS, was unmet; however, in the subgroup of patients older than 65 years, the FLO regimen achieved improved efficacy in terms of response rate, PFS, and overall survival (OS) as compared with the FLP regimen.

In a previous study, we used a modified FOLFOX regimen with the omission of bolus 5-FU with the aim to improve tolerability of such regimen in the elderly population, while preserving the outcome. This strategy was adopted based on the results of previous and ongoing studies of oxaliplatin/5-FU combination regimens. We attained an overall response rate of 34.9 %, which compared favorably with other phase II studies of FOLFOX chemotherapy, ranging from 32.2 % to 52.5 % (see Table 5). This overall response rate was noteworthy if we consider that all the patients had metastatic or recurrent gastric cancer compared with other studies in which a variable percentage (from 8 % to 35 %) of enrolled patients had locally advanced disease. We observed no grade 4 toxicity, whereas grade 1-3 gastrointestinal toxicities were reported in a moderate number of patients. The modified FOLFOX (m FOLFOX) regimen showed a 9.3% occurrence of grade 3 to 4 neutropenia, which is lower than reported in other studies.

Capecitabine monotherapy was shown an effective maintenance treatment after chemotherapy with a favorable safety profile. In metastatic breast cancer, single-agent capecitabine was administered at a dose of 1000 mg/m2 twice daily for 14 days, followed by a 7-day rest period, every 3 weeks. Short-course XELOX followed by capecitabine maintenance therapy, at a dose of 1,250 mg/m2 bid on d1-14 every 21 days until disease progression, provides an active and well-tolerated treatment option for patients with previously untreated metastatic colorectal cancer. This approach minimises the risk of unwanted cumulative neurotoxicity, is cheaper and more convenient for both patients and healthcare providers.

Recently, fixed low-dose capecitabine (1,000 mg b.i.d.), administered continuously, has been administered to patients with gastrointestinal cancers with a high level of safety. Capecitabine 1,000 mg twice daily without interruption was used for the first 11 patients. The dose was reduced to 1,000 mg twice daily 5 days per week in 8 patients who developed hand-foot syndrome. Main toxicities were grade 1 to 2 fatigue and hand-foot syndrome.

The present study is aimed to collect data on progression free survival (PFS) of elderly population with metastatic or recurrent gastric cancer, which are treated with the modified FOLFOX protocol followed by capecitabine maintenance. The aim of the present observational study is to assess if maintenance with capecitabine after a fixed number (8 cycles) of m FOLFOX regimen is able to prolong the PFS, with acceptable toxicity. In this case patients could achieve a safe treatment, sparing unnecessary combination-related toxicity (e.g. neurotoxicity, neutropenia, diarrhea and mucositis).

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients (aged ≥65 years)
2. Histologically or cytologically confirmed gastric adenocarcinoma, including gastric or gastroesophageal-junction adenocarcinoma (GEJ)
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (0-1 for patients aged ≥70 years, or with important comorbidity);
4. Measurable disease (revised RECIST) version 1.1. based on computed tomography
5. Adequate bone marrow, hepatic, and renal function, as evidenced by:
6. At least 4 weeks and recovery from effects of prior major surgery or radiation therapy
7. Ability to swallow an oral solid-dosage form of medication, including when a feeding tube is present
8. A negative serum pregnancy test within 7 days prior to accrual in women of childbearing potential (that is, all women except those who are post menopause for > 1 year or who have a history of hysterectomy or surgical sterilization)
9. Agreement to use an effective form of contraception
10. Ability to comprehend and to comply with the requirements of the study
11. Estimated life expectancy ≥3 months
12. Adequate information and subsequent written informed consent

Exclusion Criteria:

1. Previous chemotherapy for metastatic/recurrent disease, except adjuvant chemotherapy completed at least 12 months before enrollment,
2. Previous treatment with oxaliplatin
3. Squamous cell gastric carcinoma
4. Bone-only metastatic disease significant gastrointestinal bleeding ,
5. Peripheral-neuropathy > grade 2, History or presence of brain metastasis or leptomeningeal disease
6. Operable gastric or GEJ cancer
7. Herceptin (HER) 2 positive disease if the subject has not previously been treated with an anti -Herceptin (HER) 2 agent
8. Uncontrolled diarrhea, defined as more than 3 loose bowel movements above the subject's usual number of bowel movements on at least 3 days within the 14 days prior to study entry
9. Nausea or vomiting for at least 3 consecutive days within the 14 days prior to study entry despite the administration of standard antiemetic therapy
10. Known malabsorptive disorder
11. Second cancer (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the subject has been disease-free for 5 or more years)
12. Human immunodeficiency virus infection based on history of positive serology
13. Significant medical disease other than gastric cancer, including but not limited to uncontrolled diabetes mellitus, active angina or heart failure, uncontrolled hypertension, or an active psychiatric condition that would prevent consistent and compliant participation in the study
14. Presence of neuropathy > Grade 1
15. Prior radiation therapy to more than 25% of the bone marrow
16. Need for other anticancer treatment (such as chemotherapy, radiation therapy, or biologic therapy with an approved or investigational agent) while receiving protocol therapy
17. History of severe or unexpected reaction to fluoropyrimidine therapy
18. History of hypersensitivity to fluoropyrimidine agents or any of their ingredients.
19. Known dihydropyrimidine dehydrogenase deficiency
20. Pregnancy or lactation

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with recurrent or metastatic gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 6 months
  progression-free survival

SECONDARY OUTCOMES:
PFS on capecitabine maintenance | 6 months
  PFS on capecitabine maintenance
overall survival | 12 months
  overall survival
number of patients with adverse events | 12 months
  number of patients with adverse events
time to treatment failure | 12 months
  time to treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Catalano, MD, Principal Investigator — AORMN, U.O.C. Oncologia, Ospedale San Salvatore
Locations (2):
- Italy (2):
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Presidio Ospedaliero San Salvatore, Pesaro, PU
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Presidio San Salvatore,, Pesaro

REFERENCES:
- [Background] Catalano V, Bisonni R, Graziano F, Giordani P, Alessandroni P, Baldelli AM, Casadei V, Rossi D, Fedeli SL, D'Emidio S, Giustini L, Fiorentini G. A phase II study of modified FOLFOX as first-line chemotherapy for metastatic gastric cancer in elderly patients with associated diseases. Gastric Cancer. 2013 Jul;16(3):411-9. doi: 10.1007/s10120-012-0204-z. Epub 2012 Oct 11. PMID 23065042
- [Background] Catalano V, Vincenzi B, Giordani P, Graziano F, Santini D, Baldelli AM, Alessandroni P, Schiavon G, Rossi D, Casadei V, D'Emidio S, Luzi Fedeli S, Tonini G, Fiorentini G. Sequential chemotherapy with cisplatin, leucovorin, and 5-fluorouracil followed by docetaxel in previously untreated patients with metastatic gastric cancer: a phase II study. Gastric Cancer. 2012 Oct;15(4):419-26. doi: 10.1007/s10120-011-0134-1. Epub 2012 Jan 12. PMID 22237659
- [Background] De Vita F, Giuliani F, Silvestris N, Catalano G, Ciardiello F, Orditura M. Human epidermal growth factor receptor 2 (HER2) in gastric cancer: a new therapeutic target. Cancer Treat Rev. 2010 Nov;36 Suppl 3:S11-5. doi: 10.1016/S0305-7372(10)70014-1. PMID 21129604
- [Background] Catalano V, Labianca R, Beretta GD, Gatta G, de Braud F, Van Cutsem E. Gastric cancer. Crit Rev Oncol Hematol. 2009 Aug;71(2):127-64. doi: 10.1016/j.critrevonc.2009.01.004. Epub 2009 Feb 20. PMID 19230702
- See also: International group of endovascular oncology (IGEVO) website — http://igevo.jimdo.com/